CLINICAL TRIAL: NCT01330914
Title: Effects of Gastric Bypass Surgery on Calcium Metabolism and the Skeleton
Brief Title: Effects of Gastric Bypass Surgery and Calcium Metabolism and the Skeleton
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ENDB-007-10F; 1IK2CX000549-01 (NIH)
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Obesity, Morbid; Gastric Bypass
Keywords: Obesity, Morbid; Bariatric Surgery; Gastric Bypass; Calcium Metabolism Disorders; Vitamin D; Bone Density; Body Composition; Weight Loss
MeSH Terms: conditions — Obesity, Morbid; Calcium Metabolism Disorders; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gastric Bypass Surgery Patients: Obese men and women undergoing gastric bypass surgery

SUMMARY:
Obesity is a chronic illness of staggering proportions. Because weight loss through diet and exercise is difficult to attain and maintain, there has been escalating interest in bariatric surgery, including Roux-en-Y gastric bypass. Gastric bypass surgery results in long-term weight loss, dramatic improvement in comorbidities such as diabetes, and decreased mortality. Emerging evidence suggests, however, that gastric bypass may have negative effects on bone health. Because of the serious consequences of osteoporosis and fracture, this is of great concern. This study of the effects of gastric bypass on calcium metabolism and the skeleton may positively impact the clinical care of gastric bypass patients by their surgeons, primary care providers, and endocrinologists. Further, the knowledge gained may inform future investigation into the relationships between obesity, weight loss, and bone biology.

ELIGIBILITY:
Inclusion Criteria:

Scheduled to undergo gastric bypass surgery. Please note that to be eligible, one must already be working with a bariatric surgeon and with plans in place to undergo gastric bypass. This study is unable to arrange or pay for gastric bypass surgery.

Exclusion Criteria:

* Perimenopausal women
* Known intestinal malabsorption
* Prior bariatric surgery
* Use of medications known to impact bone and mineral metabolism
* Disease known to affect bone
* Illicit drug use or alcohol use >3 drinks/day
* Serum calcium >10.2 mg/dL
* Calculated creatinine clearance <30 mL/min
* Weight >350 pounds
* Wrist circumference >12 inches or calf circumference >17 inches

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women 25 to 70 years old scheduled to undergo gastric bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-07; Primary Completion 2014-04 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne L Schafer, MD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

REFERENCES:
- [Result] Schafer AL, Weaver CM, Black DM, Wheeler AL, Chang H, Szefc GV, Stewart L, Rogers SJ, Carter JT, Posselt AM, Shoback DM, Sellmeyer DE. Intestinal Calcium Absorption Decreases Dramatically After Gastric Bypass Surgery Despite Optimization of Vitamin D Status. J Bone Miner Res. 2015 Aug;30(8):1377-85. doi: 10.1002/jbmr.2467. Epub 2015 May 21. PMID 25640580
- [Result] Schafer AL, Li X, Schwartz AV, Tufts LS, Wheeler AL, Grunfeld C, Stewart L, Rogers SJ, Carter JT, Posselt AM, Black DM, Shoback DM. Changes in vertebral bone marrow fat and bone mass after gastric bypass surgery: A pilot study. Bone. 2015 May;74:140-5. doi: 10.1016/j.bone.2015.01.010. Epub 2015 Jan 17. PMID 25603463
- [Derived] Chakhtoura MT, Nakhoul NF, Akl EA, Safadi BY, Mantzoros CS, Metzendorf MI, El-Hajj Fuleihan G. Oral vitamin D supplementation for adults with obesity undergoing bariatric surgery. Cochrane Database Syst Rev. 2024 Oct 1;10(10):CD011800. doi: 10.1002/14651858.CD011800.pub2. PMID 39351881

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women and men 25-70 years of age were recruited from two academic bariatric surgery centers (the University of California, San Francisco and the San Francisco Veterans Affairs Medical Center), where surgeons used the same standardized surgical approach to Roux-en-Y gastric bypass.
Period: Overall Study
Arm/Group | Gastric Bypass Surgery Patients
Started | 55
Completed | 48
Not Completed | 7
Not completed — Withdrawal by Subject | 4
Not completed — No longer eligible (sleeve gastrectomy) | 3

BASELINE CHARACTERISTICS:
Arm/Group | Gastric Bypass Surgery Patients
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 12
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55
Menopausal status [Number; unit: participants]
  Premenopausal | 30
  Postmenopausal | 14
  N/A (Men) | 11
Weight [Mean (Standard Deviation); unit: kg] | 122.7 (19.3)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 44.2 (7.0)
Percentage body fat [Mean (Standard Deviation); unit: percentage of body fat] | 46.7 (5.9)
Diabetes status [Number; unit: participants]
  Diabetic | 22
  Not diabetic | 33
Femoral neck areal bone mineral density (DXA) [Mean (Standard Deviation); unit: g/cm2] | 0.949 (0.133)
Spine volumetric bone mineral density (QCT) [Mean (Standard Deviation); unit: g/cm3] | 0.159 (0.036)

OUTCOME MEASURES:

1. Primary Outcome: Change in Intestinal Calcium Absorption
Description: Change in fractional calcium absorption, determined by dual stable isotope method.
  Fractional calcium absorption is the fraction of ingested calcium that is absorbed, which is expressed here as the percentage of ingested calcium that is absorbed. The 6-month change is the mean difference in percentage absorption between time points. For example, if fractional calcium absorption were to decrease from 30% preoperatively to 25% at the 6-month postoperative time point, the change in fractional calcium absorption would be -5%.
Time Frame: 6 months (between baseline and 6 months)
Population: Participants from the cohort who underwent assessment of fractional calcium absorption preoperatively and 6 months postoperatively
Measure: Mean (Standard Deviation); unit: % of ingested calcium that is absorbed
Arm/Group | Gastric Bypass Surgery Patients
Number analyzed (Participants) | 33
% of ingested calcium that is absorbed | -25.8 (15.3)

2. Secondary Outcome: Areal Bone Mineral Density (BMD) at the Femoral Neck
Description: Areal BMD at the femoral neck by dual-energy X-ray absorptiometry (DXA). The 12-month change is the percentage change between the 12 month and baseline time points.
Time Frame: 12 months post-operatively (between baseline and 12 months)
Population: participants who underwent DXA at pre-op and 12-month post-op time points
Measure: Mean (Standard Deviation); unit: percent of baseline value
Arm/Group | Gastric Bypass Surgery Patients
Number analyzed (Participants) | 45
percent of baseline value | -8.0 (4.9)

3. Secondary Outcome: Trabecular Number at the Tibia
Description: Trabecular number at the tibia by high-resolution peripheral quantitative computed tomography (HR-pQCT). The 12-month change is the percentage change between the 12 month and baseline time points. HR-pQCT images were analyzed using the manufacturer's standard clinical evaluation protocol, with trabecular structure extracted using a threshold-based binarization process.
Time Frame: 12 months post-operatively (between baseline and 12 months)
Population: participants who underwent HR-pQCT at pre-op and 12-month post-op time points
Measure: Mean (Standard Deviation); unit: percent of baseline value
Arm/Group | Gastric Bypass Surgery Patients
Number analyzed (Participants) | 44
percent of baseline value | -4.6 (8.4)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Participants were asked about interim adverse events at baseline, 6-month, and 12-month study visits. Adverse events volunteered by participants between study visits were also recorded.
Arm/Group | Gastric Bypass Surgery Patients
Serious Adverse Events (participants affected / at risk) | 1/55
Other Adverse Events (participants affected / at risk) | 3/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gastric Bypass Surgery Patients (N=55)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.82% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gastric Bypass Surgery Patients (N=55)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No